CLINICAL TRIAL: NCT06909188
Title: The Study of Association of Helicobacter Infections in Biliary Tract Cancers
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS- BILIARY TRACT CANCERS01
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Histopathology Samples will be assessed for immuno histochemistry and Polymerase chain reaction for Helicobacter species identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Benign Gallbladder diseases: Patients with Benign biliary disease(Gall stone disease) undergoing laparoscopic cholecystectomy will be included
  Interventions: Other: No intervention
- Voluntary healthy liver donors: Gall bladder samples from Voluntary Healthy liver donors undergoing cholecystectomy.
  Interventions: Other: No intervention
- Patients with high risk for biliary tract malignancy: Choledochal cyst Porcelain Gallbladder Gallbladder polyp Primary sclerosing cholangitis Metaplasia / dysplasia Stone size >2 cm Abnormal pancreaticobiliary duodenal junction(APBDJ) Cholecystectomy in patients with both Hepatitis B and C Cholecystectomy in age more than 60 years Hepaticolithiasis
  Interventions: Other: No intervention
- Biliary tract carcinoma: Patients undergoing surgery for biliary tract cancers.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
Biliary tract carcinoma (BTC) includes gallbladder carcinoma, hilar cholangiocarcinoma, and distal cholangiocarcinoma, intrahepatic cholangiocarcinoma. Chronic infections of the biliary tract are major drivers of cancer. Helicobacter species is one of the most established pro-oncogenic pathogens for gastric malignancy.

In addition to H Pylori, H.bilis and H.hepaticus have a significantly higher incidence in bile from biliary tract and gallbladder cancer patients than in patients with gallstones/cholecystitis.

This, together with the high prevalence of gallstones, makes it important to evaluate the role of Helicobacter in biliary tract cancers. This study aims to compare the prevalence of Helicobacter sp.(pylori, bilis, hepaticus). This study will include biliary tract carcinoma patients, benign biliary disease patients, high risk conditions for malignancy and Voluntary healthy liver donors with no gallbladder pathology. HPE samples will be assessed and association of Helicobacter sp will be studied among all 4 arms.

All the included samples will be assessed for Helicobacter species using giemsa stain and DNA PCR. Results will be studied to compare the prevalence of Helicobacter sp. in Biliary tract malignancy and benign biliary diseases.

DETAILED DESCRIPTION:
Biliary tract carcinoma (BTC) includes gallbladder carcinoma, hilar cholangiocarcinoma, and distal cholangiocarcinoma, intrahepatic cholangiocarcinoma. Chronic infections of the biliary tract are major drivers of cancer. Helicobacter species is one of the most established pro-oncogenic pathogens for gastric malignancy. However, its role in biliary tract cancers is under investigation. Recently H. pylori has been associated with gallbladder pathologies like cholelithiasis, cholecystitis, choledocholithiasis, gallbladder polyps. However, some studies have also reported that chronic inflammation due to H. pylori infection causes biliary tract cancer. On the other hand, some studies have reported no association between H. pylori infection and gallbladder diseases. In addition to H Pylori, H.bilis and H.hepaticus have a significantly higher incidence in bile from biliary tract and gallbladder cancer patients than in patients with gallstones/cholecystitis.This, together with the high prevalence of gallstones, makes it important to evaluate the role of Helicobacter in biliary tract cancers. This study aims to compare the prevalence of Helicobacter sp.(pylori, bilis, hepaticus). This study will include biliary tract carcinoma patients, benign biliary disease patients, high risk conditions for malignancy and Voluntary healthy liver donors with no gallbladder pathology. HPE samples will be assessed and association of Helicobacter sp will be studied among all 4 arms. Patients who have received H pylori eradication therapy will be excluded. All the included samples will be assessed for Helicobacter species using giemsa stain and DNA PCR. Results will be studied to compare the prevalence of Helicobacter sp. in Biliary tract malignancy and benign biliary diseases.

ELIGIBILITY:
Inclusion Criteria:

* Biliary tract carcinoma patients who underwent resection
* Patients undergoing cholecystectomy for benign biliary disease.
* Voluntary healthy liver donors with no gallbladder pathology
* Patients undergoing cholecystectomy for conditions with high risk of malignancy

Exclusion Criteria:

* Patients who have taken H.pylori eradication previously in last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biliary tract carcinoma patients , Benign biliary disease undergoing laparoscopic cholecystectomy Healthy donors without any GB pathology and Retrospective samples of high risk/ precursor biliary condition.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To compare the prevalence of Helicobacter sp. in Biliary tract cancers and benign biliary diseases. | day 0

SECONDARY OUTCOMES:
To assess correlation of Helicobacter infection with disease stage in Biliary tract cancers. | day 0
To assess the correlation of Helicobacter infection with high risk conditions - | day 0

CONTACTS AND LOCATIONS:
Locations (1):
- ILBS, New Delhi, National Capital Territory of Delhi, India